CLINICAL TRIAL: NCT01795742
Title: Equivalence of a Human-Powered Nebulizer to an Electric Nebulizer in the Treatment of Mild to Moderate Asthma in El Salvador
Brief Title: Equivalence of a Human-Powered Nebulizer to an Electric Nebulizer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marquette University (Other)
Responsible Party: Principal Investigator, Lars Olson, Associate Professor of Biomedical Engineering, Marquette University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MU-HR-2433
Record Dates: First submitted 2013-02-03; First posted 2013-02-21 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Asthma
Keywords: Asthma; Nebulizers; Salbutamol; Developing Countries
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electric Nebulizer (Active Comparator): Pulmo-Aide Model 5650D
  Interventions: Device: Human-Powered Nebulizer
- Human-Powered Nebulizer (Experimental): Human-Powered
  Interventions: Device: Human-Powered Nebulizer

INTERVENTIONS:
Device: Human-Powered Nebulizer

SUMMARY:
This is an equivalence study comparing an electric nebulizer with a human-powered nebulizer--one that does not need electricity--in the treatment of mild to moderate asthma exacerbations in a regional clinic in San Salvador, El Salvador.

DETAILED DESCRIPTION:
The study design is to treat individuals suffering from mild to moderate exacerbations of asthma with nebulized salbutamol (2.5mg). Subjects will receive nebulization using either an electric nebulizer compressor or a human-powered nebulizer compressor. Improvement in peak expiratory flow will be the primary endpoint. Blood oxygenation levels as measured by pulse oximetry will be a secondary endpoint of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from Mild or Moderate Asthma symptoms
* Increased respiratory rate, but not over 30 breaths per minute
* Reduced peak expiratory flow rate, but not less than 60% of normal
* Oxygen saturation levels reduced but greater than 90%

Exclusion Criteria:

* Any other respiratory condition that would interfere with nebulizer treatment
* If any other medication is being taken at the time
* Pregnant women or women who may think they might be pregnant
* Never taken salbutamol before

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2012-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Improvement in Peak Expiratory Flow | From before to after nebulizer treatment lasting approximately 30 minutes

SECONDARY OUTCOMES:
Improvement in blood oxygenation as measured by pulse oximetry | From before to after nebulizer treatment lasting about 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Lars E Olson, Ph.D., Principal Investigator — Marquette University
Locations (1):
- Hospital Nacional San Bartolo, Ilopango, San Salvador Department, El Salvador

REFERENCES:
- [Derived] Hallberg CJ, Lysaught MT, Najarro RA, Cea Gil F, Villatoro C, Diaz de Uriarte AC, Olson LE. Treatment of asthma exacerbations with the human-powered nebuliser: a randomised parallel-group clinical trial. NPJ Prim Care Respir Med. 2014 Jun 26;24:14016. doi: 10.1038/npjpcrm.2014.16. PMID 24965834